CLINICAL TRIAL: NCT06407648
Title: Using Personalized Assessments in the Treatment of Childhood OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00406231
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: children; adolescents; exposure with response prevention; cognitive behavioral therapy; ERP; CBT
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized parallel clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Assessments (Experimental): 12 sessions of exposure with response prevention (ERP) that is guided by personalized assessments.
  Interventions: Other: Personalized Assessments
- Standard of Care (Active Comparator): 12 sessions of exposure with response prevention (ERP) that is guided using standard practice.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Personalized Assessments — Personalized CBT will use individualized OCD symptom networks to guide CBT strategies to target central symptom nodes in contemporaneous networks.
  Arms: Personalized Assessments
Other: Standard of Care — The standard CBT condition will use standard-of-care approaches to guide CBT strategies to target OCD symptoms.
  Arms: Standard of Care

SUMMARY:
The primary purpose of this study is to learn whether personalized assessment of obsessive-compulsive disorder (OCD) symptoms in childhood OCD using mobile health technology are feasible and acceptable for youth and parents. The investigators will also examine whether personalized cognitive-behavioral therapy (CBT) that is informed by personalized OCD assessments yields better clinical outcomes when compared to standard CBT for youth with OCD

ELIGIBILITY:
Inclusion Criteria:

1. be 8-17 years of age;
2. meet diagnostic criteria for a primary diagnosis of OCD on a structured clinical interview;
3. have moderate OCD severity as evidenced by a CY-BOCS total score of ≥16;
4. medication free and/or on a stable dose of medication 8 weeks prior to study participation;
5. be English speaking.

Exclusion Criteria:

1. the presence of psychotic disorder, bipolar disorder, or autism spectrum disorders;
2. significant suicidal ideation that warrants medical intervention;
3. concurrent psychotherapy for OCD;
4. inability to complete scales, or attend visits.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale Second Edition (CY-BOCS-II) Total Severity Score | Screen, Baseline (Week 0), Week 4, Week 8, and Week 12
  A clinician-rated measure of OCD symptom severity in the past week. This 10-item measure is rated on a 0 to 5 scale with a total score ranging from 0 to 50. A higher total score is reflective of greater OCD symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. McGuire, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No